CLINICAL TRIAL: NCT07318272
Title: Comparison of Clinical and Functional Outcomes After Anterior Cruciate Ligament Reconstruction and Primary Repair Surgery
Brief Title: Clinical and Functional Outcomes After ACL Reconstruction Versus Primary Repair
Status: Not yet recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Dudu Özdemir, MSc., Gazi University
Other Study IDs: Gazi2025
Record Dates: First submitted 2025-12-08; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament (ACL) Tear; Anterior Cruciate Ligament Reconstruction; Isokinetic Test
Keywords: ACL Injury; Anterior Cruciate Ligament; ACL Reconstruction; ACL Primary Repair; Postoperative Outcomes; Muscle Oxygenation; Isokinetic Testing
MeSH Terms: conditions — Lacerations; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ACL Reconstruction Group: Demographic data, injury history, and surgical details will be recorded for all participants. The International Physical Activity Questionnaire, IKDC, and ACL-RSI scales will be administered. Assessments will be completed over two days. Isokinetic knee flexor/extensor strength, fatigue protocol, and H/Q ratios will be measured using the Cybex Norm dynamometer. Quadriceps and hamstring muscle oxygenation will be assessed with Train.Red NIRS. Knee proprioception will be evaluated via active joint repositioning, and postural control and dynamic stability will be measured using the KFORCE force platform. Knee laxity will be assessed with the GNRB arthrometer.
- Primary ACL Repair Group: Demographic data, injury history, and surgical details will be recorded for all participants. The International Physical Activity Questionnaire, IKDC, and ACL-RSI scales will be administered. Assessments will be completed over two days. Isokinetic knee flexor/extensor strength, fatigue protocol, and H/Q ratios will be measured using the Cybex Norm dynamometer. Quadriceps and hamstring muscle oxygenation will be assessed with Train.Red NIRS. Knee proprioception will be evaluated via active joint repositioning, and postural control and dynamic stability will be measured using the KFORCE force platform. Knee laxity will be assessed with the GNRB arthrometer.
- Healthy Control Group: Demographic data and physical activity levels will be recorded for healthy participants. All individuals will complete the International Physical Activity Questionnaire, IKDC, and ACL-RSI scales. Assessments will be conducted over two days. Knee flexor/extensor strength and H/Q ratios will be measured using the Cybex Norm isokinetic dynamometer. Quadriceps and hamstring muscle oxygenation will be assessed with the Train.Red NIRS device. Knee proprioception will be measured using an active joint repositioning test, while postural control and dynamic stability will be evaluated with the KFORCE force platform. Knee laxity will be assessed using the GNRB arthrometer.

SUMMARY:
The anterior cruciate ligament (ACL) is the primary structure responsible for controlling anterior-posterior translation and rotational stability of the knee joint. Although ACL reconstruction has long been considered the gold standard among surgical interventions following ACL injury, arthroscopic primary repair techniques have recently regained interest. With advances in minimally invasive surgical procedures, refined patient selection criteria, and improved rehabilitation strategies, the clinical effectiveness of primary repair is once again being re-evaluated. However, there remains a limited body of literature directly comparing the medium- to long-term effects of these two surgical techniques on neuromuscular performance, fatigue tolerance, and functional outcomes.

The aim of this study is to comparatively investigate postoperative muscle strength and endurance, isokinetic fatigue response, muscle oxygenation, proprioception, knee stability, postural control, and patient-reported outcome measures in individuals who have undergone ACL reconstruction or primary repair. Assessments will include low- and high-velocity tests performed on the Cybex Norm isokinetic dynamometer, a 33-repetition fatigue protocol at 300°/s, muscle oxygenation analysis using Train.Red NIRS, knee laxity measurement via the GNRB arthrometer, single-leg balance and landing evaluations using the KFORCE force platform, and subjective outcome measures (IKDC, ACL-RSI).

The findings of this study are expected to provide a more comprehensive understanding of how surgical technique influences physiological, biomechanical, and functional outcomes. This knowledge may contribute to the development of individualized rehabilitation approaches and evidence-based return-to-sport criteria.

DETAILED DESCRIPTION:
The anterior cruciate ligament (ACL), one of the key stabilizers of the knee joint, plays a crucial role in maintaining both anteroposterior and rotational stability. The increasing popularity of recreational and competitive sports has contributed to a rising incidence of ACL injuries in recent years. Until the late 1980s, primary repair was widely accepted as the standard treatment for ACL injuries. Although short-term outcomes were generally satisfactory, this technique was largely abandoned due to high failure rates observed in medium- and long-term follow-ups. The probable causes of these unfavorable outcomes include suboptimal patient selection, invasive open repair techniques performed with absorbable sutures, and nonfunctional rehabilitation approaches characterized by prolonged cast immobilization. Considering the limited healing potential of the ligament, reconstruction surgery-performed using allografts or autologous tendon grafts-emerged as the new standard for the treatment of ACL injuries.

However, several disadvantages associated with reconstruction have raised the notion that a single surgical method may not be appropriate for all patients. These drawbacks include graft rerupture or contralateral ACL injury, loss of proprioception, physeal disturbances in pediatric populations, donor site morbidity in autografts or higher failure rates in allografts, the potential need for complex revision surgery, and the risk of early-onset osteoarthritis. In recent years, advances in patient selection criteria, minimally invasive surgical techniques, and modern rehabilitation protocols have renewed interest in arthroscopic primary ACL repair. This method preserves the native ligament and its proprioceptive properties while avoiding donor site morbidity, thereby offering the potential for a smoother and more accelerated postoperative rehabilitation process. Additionally, if primary repair fails, ACL reconstruction remains a viable subsequent treatment option. Primary repair has been described as a less morbid surgical alternative for patients presenting with acute proximal ACL tears, although high-quality evidence for its use is still limited.

Recent studies have shown improved success rates following primary repair of proximal ACL tears. In one investigation, researchers reported a 0% failure rate among 75 patients treated with primary ACL repair. Furthermore, 88% of patients demonstrated a negative pivot-shift test, 87% exhibited 0 or +1 Lachman test findings, and 89% successfully returned to sport. Similarly, numerous studies have evaluated the clinical effectiveness of ACL repair, and several recent systematic reviews have suggested that primary repair may be an effective treatment strategy with reasonable clinical outcomes compared to ACL reconstruction. Nonetheless, concerns remain that some evidence includes older cohorts that may not reflect contemporary surgical practices. A systematic review of only five comparative studies found no significant differences between treatments regarding clinical outcome scores, knee laxity, or graft rerupture rates. More recent randomized controlled trials have yielded conflicting results; some authors report that ACL repair provides non-inferior clinical outcomes compared to reconstruction, while others emphasize higher rates of adverse events and failure associated with repair. These issues underscore the need for further research comparing the medium- to long-term outcomes of ACL repair and ACL reconstruction.

Given the recent increase in clinical studies evaluating ACL repair versus reconstruction, synthesizing and expanding evidence from such research is critical for achieving a comprehensive and transparent understanding of the advantages, disadvantages, and clinical implications of both procedures.

The purpose of the present study is to compare postoperative clinical outcomes and patient-reported measures in individuals undergoing ACL reconstruction or primary ACL repair. Long-term outcomes of both procedures will be examined in terms of knee flexor and extensor muscle strength and endurance, torque-generating capacity and fatigue resistance, muscle oxygenation, knee joint proprioception, lower-extremity balance, and knee laxity. In this context, the findings of this study aim to provide valuable insights that may inform postoperative rehabilitation strategies and contribute to evidence-based clinical decision-making.

ELIGIBILITY:
Inclusion Criteria for the ACL Reconstruction Group

* Age 18-40 years
* History of complete ACL rupture treated with ACL reconstruction
* Surgery performed at Gazi University Department of Orthopedics and Traumatology
* At least 12 months postoperative at the time of evaluation
* Ability to comply with all study procedures
* Signed informed consent

Exclusion Criteria for the ACL Reconstruction Group

* Previous surgery for partial or chronic ACL tear
* Concomitant multi-ligament knee injuries
* Prior surgery on the ipsilateral or contralateral knee
* Lower extremity malalignment (e.g., significant varus/valgus)
* Tibial avulsion-type ACL injury
* Neurological or musculoskeletal disorders affecting lower limb function
* Any medical condition that may interfere with test performance or safety

Inclusion Criteria for the Primary ACL Repair Group

* Age 18-40 years
* Complete ACL rupture treated with arthroscopic primary ACL repair
* Surgery performed at Gazi University Department of Orthopedics and Traumatology
* Minimum 12 months postoperative at the time of assessment A-bility to follow and complete study procedures
* Signed informed consent

Exclusion Criteria for the Primary ACL Repair Group

* Previous surgery for partial or chronic ACL injury
* Multi-ligament knee injuries
* History of surgery on either knee
* Lower extremity malalignment
* Tibial avulsion-type ACL rupture
* Neuromuscular or musculoskeletal diseases affecting lower limb function or balance
* Any condition that may affect participation or compromise safety

Inclusion Criteria for the Healthy Control Group

* Age 18-40 years
* No significant lower-extremity malalignment (e.g., varus/valgus deformity)
* No history of lower-extremity injury within the past 12 months
* No known chronic systemic disease
* No history of knee surgery or diagnosed knee pathology
* Ability to understand and comply with study procedures
* Signed informed consent

Exclusion Criteria for the Healthy Control Group

* Presence of clinically significant lower-extremity malalignment
* Lower-extremity musculoskeletal injury within the last 12 months
* Any chronic systemic or metabolic disease
* History of knee injury, knee surgery, or diagnosed knee pathology
* Neurological, vestibular, or musculoskeletal disorder affecting balance or gait
* Inability to complete study procedures

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include a total of 45 participants. All participants will be adults aged 18-40 who meet the study's eligibility criteria, are able to comply with the assessment procedures, and provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Peak Torque (Isokinetic Strength) | First Day
  Peak torque of the knee flexor and extensor muscles will be measured using an isokinetic dynamometer (Cybex NORM® isokinetic dynamometer, Humac, CA, USA). Measurements will be performed in the following modes: concentric contraction at 60°/s, eccentric contraction at 60°/s, concentric contraction at 180°/s, and concentric contraction at 300°/s. Peak torque values will be recorded for each testing velocity and contraction mode and expressed in Newton-meters (Nm).
  Unit of Measure: Newton-meter (Nm)
Extremity Symmetry Index (ESI) | First day
  Extremity Symmetry Index will be calculated by comparing the involved and uninvolved limbs using peak torque values obtained from isokinetic testing.
  Unit of Measure: Percentage (%)
Conventional Hamstring-to-Quadriceps Ratio (H/Q Ratio) | First day
  The conventional H/Q ratio will be calculated as the ratio of concentric hamstring peak torque to concentric quadriceps peak torque. Unit of Measure: Ratio
Functional Hamstring-to-Quadriceps Ratio | First day
  The functional H/Q ratio will be calculated as the ratio of eccentric hamstring peak torque to concentric quadriceps peak torque. Unit of Measure: Ratio
Functional Range | First Day
  Functional range will be defined as the angular range in which at least 85% of peak torque is maintained during isokinetic testing. Unit of Measure: Percentage (%)
Fatigue-Induced Peak Torque Decline | First Day
  Fatigue-related performance decline will be calculated as the percentage decrease in peak torque following a 33-repetition isokinetic fatigue protocol at 300°/s. Unit of Measure: Percentage (%)
Muscle Oxygenation | First Day
  Muscle oxygenation will be assessed using the Train.Red FYER wireless near-infrared spectroscopy (NIRS) system (Train.Red, Gelderland, Netherlands). The device provides continuous, non-invasive measurements of tissue oxygen saturation (StO₂) and the oxy-deoxyhemoglobin difference (HbDiff). Sensors will be placed over the quadriceps and hamstring muscles following SENIAM guidelines. Muscle oxygenation will be recorded before and immediately after the isokinetic fatigue protocol to evaluate changes in local oxygen utilization and metabolic stress.

SECONDARY OUTCOMES:
Knee Joint Proprioception | First Day
  Knee proprioception will be assessed using an active joint repositioning test performed on the Cybex NORM® isokinetic system (Humac, CA, USA). Participants will actively reproduce a target angle (30° knee flexion) starting from 90° flexion. Three trials will be recorded, and the absolute angular error will be calculated as the mean difference between the target angle and the reproduced angles. This measure reflects the accuracy of joint position sense and will be used to evaluate proprioceptive function.
Single Leg Balance | Second Day
  Postural control will be assessed using the KFORCE Plates force platform (Kinvent, Montpellier, France). Participants will perform a single-leg balance task, and Center of Pressure (CoP)-based variables such as mean CoP velocity, path length, sway area, and stabilization time will be recorded. Measurements will be obtained under standardized testing conditions for both limbs.
Single Leg Landing | Second Day
  Dynamic stability will be assessed using the KFORCE Plates force platform. Participants will perform a single-leg landing task, and Center of Pressure (CoP)-based variables including stabilization time, CoP displacement, sway area, and CoP velocity will be analyzed. This measure evaluates the participant's ability to achieve stable posture following landing.
Knee Laxity | First Day
  Knee anterior laxity will be assessed using the GNRB® arthrometer at 20° of knee flexion. The primary outcome variable will be Anterior Tibial Translation (ATT) measured in millimeters under standardized forces (134 N and 200 N). The side-to-side difference in ATT and the slope value (stiffness index) will also be recorded to evaluate anterior cruciate ligament integrity. These parameters provide an objective and quantitative measure of ligamentous stability.
IKDC Subjective Knee Evaluation | First Day
  The International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form will be used to assess patient-reported knee symptoms, function, and sports activity levels. Scores range from 0 to 100, with higher scores indicating better knee function and fewer symptoms. This measure provides a validated assessment of functional recovery following ACL surgery.
ACL-RSI (Return to Sport Index) | First Day
  The Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) scale will be administered to evaluate psychological readiness to return to sport. The 12-item scale assesses emotions, confidence, and risk appraisal related to returning to physical activity. Scores range from 0 to 100, with higher scores indicating greater psychological readiness. This measure allows comparison of psychological recovery after ACL reconstruction and primary repair.

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Karatas, Prof. Dr., Study Director — Gazi University; Dudu Ozdemir Can, MSc, Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoogeslag RAG, Brouwer RW, Boer BC, de Vries AJ, Huis In 't Veld R. Acute Anterior Cruciate Ligament Rupture: Repair or Reconstruction? Two-Year Results of a Randomized Controlled Clinical Trial. Am J Sports Med. 2019 Mar;47(3):567-577. doi: 10.1177/0363546519825878. PMID 30822124
- [Background] Szwedowski D, Paczesny L, Zabrzynski J, Gagat M, Domzalski M, Huri G, Widuchowski W. The Comparison of Clinical Result between Primary Repair of the Anterior Cruciate Ligament with Additional Internal Bracing and Anatomic Single Bundle Reconstruction-A Retrospective Study. J Clin Med. 2021 Aug 31;10(17):3948. doi: 10.3390/jcm10173948. PMID 34501400
- [Background] Kunze KN, Pareek A, Nwachukwu BU, Ranawat AS, Pearle AD, Kelly BT, Allen AA, Williams RJ 3rd. Clinical Results of Primary Repair Versus Reconstruction of the Anterior Cruciate Ligament: A Systematic Review and Meta-analysis of Contemporary Trials. Orthop J Sports Med. 2024 Jun 11;12(6):23259671241253591. doi: 10.1177/23259671241253591. eCollection 2024 Jun. PMID 38867918
- [Background] Vermeijden HD, van der List JP, O'Brien R, DiFelice GS. Patients Forget About Their Operated Knee More Following Arthroscopic Primary Repair of the Anterior Cruciate Ligament Than Following Reconstruction. Arthroscopy. 2020 Mar;36(3):797-804. doi: 10.1016/j.arthro.2019.09.041. Epub 2020 Jan 7. PMID 31919026
- [Result] Schneider KN, Schliemann B, Gosheger G, Theil C, Weller J, Buddhdev PK, Ahlbaumer G. Good to Excellent Functional Short-Term Outcome and Low Revision Rates Following Primary Anterior Cruciate Ligament Repair Using Suture Augmentation. J Clin Med. 2020 Sep 23;9(10):3068. doi: 10.3390/jcm9103068. PMID 32977649
- [Result] Duong JKH, Bolton C, Murphy GT, Fritsch BA. Anterior cruciate ligament repair versus reconstruction: A clinical, MRI and patient-reported outcome comparison. Knee. 2023 Dec;45:100-109. doi: 10.1016/j.knee.2023.09.008. Epub 2023 Nov 3. PMID 37925800
- [Result] Ciceklidag M, Kaya I, Ayanoglu T, Ayas IH, Ozer M, Ataoglu MB, Kanatli U. Proprioception After Primary Repair of the Anterior Cruciate Ligament. Am J Sports Med. 2024 Apr;52(5):1199-1208. doi: 10.1177/03635465241228839. Epub 2024 Mar 4. PMID 38557260